CLINICAL TRIAL: NCT03498469
Title: Keeping Children in Healthy and Protective Families: Effects of a Household-based Parenting Program on Reintegration of Children Into Family-based Care in Uganda
Brief Title: Reintegration of Children Into Family-based Care in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 170901
Record Dates: First submitted 2017-12-08; First posted 2018-04-13 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Parenting
Keywords: reintegration, reunification, child development

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either of the two arms in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Randomized assignment will be done by the individuals who are evaluating the study outcomes, but will be blind to participant assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Parenting program (Active Comparator): Participants assigned to this comparison arm will receive a standardized reintegration package that includes individualized case management support and a reunification cash grant. Individualized case management will consist of a caseworker-developed individualized care plan with routine caseworker visits at the household level. At a minimum, each family will be visited on a monthly basis during the first 6 months post-placement and then every other month for the next 9 months. For the cash grant, the family of each enrolled child will receive a reunification cash grant in the Ugandan Shilling equivalent of $125, administered in two equal disbursements. It is designed to offset the cost of child care.
  Interventions: Behavioral: Standardized reintegration package
- Parenting program (Experimental): Those in the intervention arm will receive an enhanced reintegration package of services that consist of the standard package (case management and cash grant) plus a parenting program called 'Esanyu Mu Maka' or Happiness in the Home. The parenting curriculum used will be an adaptation of the evidence-based Sinovuyo Kids curriculum, tailored for caregivers of children age 1 to 13 years. It will have specifically designed components to address parenting challenges under reunification/reintegration conditions and to support the child and caregiver in building their relationship. It will be delivered at the household level by project trained parenting facilitators. The program will consist of approximately 13 bi-weekly sessions, which will be delivered over the course of 7 months.
  Interventions: Behavioral: Enhanced reintegration package

INTERVENTIONS:
Behavioral: Standardized reintegration package — Participants assigned to this comparison arm will receive a standardized reintegration package that includes individualized case management support and a reunification cash grant Individualized case management will consist of a caseworker-developed individualized care plan with routine caseworker visits at the household level. Home visitation will begin during the family assessment and preparation stages and continue throughout the 15-month post-reunification follow-up period. For the cash grant, the family of each enrolled child will receive a reunification cash grant in the Ugandan Shilling equivalent of $125, administered in two equal disbursements. It is designed to offset the cost of child care.
  Arms: No Parenting program
Behavioral: Enhanced reintegration package — Participants assigned to this arm will receive an enhanced reintegration package that consists of the parenting program, individualized case management, and the reunification grant. will be delivered at the household level by project trained parenting facilitators. The program will consist of approximately 13 bi-weekly sessions, which will be delivered over the course of 7 months. The individualized case management and the reunification grant will be similar to those in the comparison arm.
  Other Names: 'Esanyu Mu Maka' or Happiness in the Home
  Arms: Parenting program

SUMMARY:
The proposed study will be an individually randomized controlled trial with children (age 1 to 13 years at the time of screening for inclusion in the study) living in residential care, reintegrated back into family-based care, in Uganda. It is designed to evaluate the impact of adding a household-based parenting program to a standardized reintegration package that includes individualized case management support and a reunification cash grant, aimed at improving the reintegration of children living in residential care back into family-based care. The study population will include children living in residential care facilities (RCFs) in Mpigi, Mukono, Masaka and Greater Masaka districts in Uganda.

Study participants will be randomized to one of two arms of the study: the comparison arm and the intervention arm. The target sample size is 640 children with 320 in each arm of the study. Children assigned to the comparison arm will receive a standard reintegration package that includes individualized case management support and a reunification cash grant. Those in the intervention arm will receive the enhanced reintegration package that includes individualized case management support, reunification cash grant and a parenting intervention. Data will be collected at baseline (while the child is still living in the RCF), 6 months post-placement and 12 months post-placement.

Data will be collected in the local language by a project trained local data collection partner on the following six domains of reintegration: Child health and development, Psychosocial health and wellbeing of the child and primary caregiver, Protection and safety of the child, Caregiver-child relationship, Child's and caregiver's sense of social and community belonging, Education access, quality, and achievement (where age-appropriate).

The sources of data are a) interviews with primary caregiver, b) interviews with RCF caregiver, c) interviews with older children (8-13 years of age), d) standardized assessments of child cognitive functioning for all the study children, and e) focus groups and interviews with participants, parenting facilitators, and case managers.

DETAILED DESCRIPTION:
Background:

There is an expanding global evidence base that illustrates the negative effects of placement in residential care on the physical, cognitive and socioemotional development of children (Smyke, 2007). Based on this evidence, legal and policy frameworks and programming have focused on reducing reliance on residential care and strengthening family-based environments for children (United Nations General Assembly, 2009). Recent care reform initiatives in Uganda promote the reunification and reintegration of children living in RCFs back into family-based care. Reintegration encompasses more than just the relocation of separated children into family-based care; it includes multiple dimensions of children's and families' wellbeing over time.

Uganda's population is young and vulnerable, with as many as 80 to 90 percent of children living in RCFs have at least one living parent (Rotabi, 2016). In Uganda, a study by Walakira, Ddumba-Nyanzi, & Bukenya (2015) found that more than two-thirds of the children living in 28 RCFs had at least one living parent and many more had a contactable relative. Children enter residential care for a variety of reasons and while poverty is often a driving factor, other factors such as inadequate access to quality education, health care, or social services, disability, child behavior problems, parental alcohol or drug abuse and death of one or more caregiver, may also be contributing or precipitating factors.

There have been several studies that have shown beneficial effects of parenting interventions on child cognitive outcomes in Uganda (e.g., Boivin et al., 2013). A recent systematic review of 12 randomized controlled trials (RCT) examining parenting inventions in low and middle income countries found evidence that parenting interventions positively affected a range of outcomes, including parent-child interactions, parental knowledge and attitudes, and reduced self-reported harsh or abusive parenting. The authors concluded that parenting interventions "hold some promise for improving parenting practices and reducing risk factors for child maltreatment in low and middle-income countries" (Knerr et al., 2013).

Study Rationale:

While there is a growing interest and emphasis in finding ways to transition children from residential care to family-based care, there is very little rigorous evidence that identifies specific interventions that help to facilitate this process, especially within sub-Saharan Africa. The proposed study aims to contribute to the evidence base by determining whether provision of a household-based parenting program contributes to reintegration success in Uganda. The six 'domains' of reintegration success are based on the following outcomes:

1. Child Health and Development Child

   a. Child anthropometry including height, weight, BMI; access to food and health care; child cognitive development; protective factors and resilience (only for older children)
2. Psychosocial Health and Wellbeing:

   1. Child internalizing and externalizing behaviors; self-esteem (only for older children); child depressive symptoms (only for older children);
   2. Caregiver's self-esteem; symptoms of mental disorders; quality of marriage; parental stress; loneliness
3. Child Protection and Safety

   1. Child attitudes towards physical punishment (only for older children); experiences of physical, emotional, sexual abuse, and neglect (only for older children)
   2. Caregiver attitudes towards physical punishment; experiences of physical, emotional, sexual abuse, and neglect
4. Caregiver-Child Relationship

   a. Caregiver's involvement, monitoring and supervision of the child; caregiver's parenting behaviors; disturbances in attachment in young children; parent-child activity scale
5. Social and Community Belonging

   1. Child's social support (only for older children); sense of community belonging (only for older children)
   2. Caregiver's social support; sense of community belonging
6. Education Access, Quality, and Achievement

   1. Child's school enrollment, attendance, progression, and grades (if feasible);
   2. Child's satisfaction and happiness with school (only for older children

Study Partners:

The study is part of the Coordinating Comprehensive Care for Children (4Children), which is a five-year United States Agency for International Development (USAID)-funded consortium of organizations led by Catholic Relief Services (CRS) with partners IntraHealth, Maestral, Pact, Plan International, and Westat. 4Children is designed to improve health and wellbeing outcomes for orphans and vulnerable children (OVC). 4Children's Keeping Children in Healthy and Protective Families (KCHPF) project is supported by the Displaced Children and Orphans Fund (DCOF). It focuses on strengthening family care among households where there is a high risk of child separation, or where children can be reintegrated into family-based care after having been placed in residential care. Westat is leading the data collection effort, in close collaboration with our partner, the Department of Social Work and Social Administration at Makerere University, which will serve as the local research partner. Westat also lead protocol development and will be responsible for sampling, data management, data analysis, and preparation of the final report and publication. The study protocol was approved by Mildmay, on May 17th, 2017.

Site Selection:

All RCFs known to district authorities in the districts of Greater Masaka, Mpigi, and Mukono were evaluated for inclusion in the study. These three districts were selected for the study given their proximity to Kampala and the fact that these districts do not have currently active, externally-funded family reintegration programs. Additionally, the Ministry of Gender, Labor and Social Development (MGLSD) and the authorities in these districts (including the Probation and Social Welfare Officers [PSWOs]) have indicated their support of the KCHPF project.

Enrollment Procedures:

A team of case managers affiliated with the KCHPF project will review the child records at each of the participating RCFs and complete bio-data forms on all of the children. This form will include information on the child's background, identity of the child's birth family or next of kin, as well as the family's location, circumstances and ability to be reunified with the child. Using this information, the case managers will conduct a rapid assessment that will allow KCHPF team to determine which children are potentially eligible for inclusion, pending further follow up with and assessment of the family. The information, aggregated over the RCFs, will be sent to Westat to help plan sample selection and randomization. Case managers will conduct family tracing efforts on potentially eligible children to assess the family's capacity and suitability for reunification. Those who meet the eligibility criteria and agree to being reunified by the KCHPF project will be included in the sampling frame.

All enrolled child-caregiver pairs will be randomized to the comparison or intervention arms of the study. The components of the reintegration packages provided in each arms are described below.

'Esanyu Mu Maka' will be delivered on a household level. The primary caregiver will be required to attend all sessions. In addition, all adults who participate in caring for the reintegrated child and ensuring her/his wellbeing will be invited to participate in the program. This will include neighbors if the neighbors also share in the caregiving of the child. Each visit will be about an hour long and will be participatory with discussions regarding home practice activities during the previous week, working through illustrated stories together, role-playing new parenting skills, and assignment of home practice for the following session. Caregiver and family participation in the parenting sessions will be documented in the parenting M&E system and may be used in the analysis. The 'Esanyu Mu Maka' curriculum will cover the list of topic shown below. However, given the broad age range of children being reintegrated (1 to 13 years), the curriculum will be customized to address the specific needs of caregivers of children 1 to 3 years, 4 to 7 years, and 8 to 13 years.

The qualitative data component will provide additional contextual data on the satisfaction and feasibility of the intervention components for children and caregivers as well as the program implementers (parenting facilitators and case managers), and the effect of the individual intervention components on the reintegration process from the perspectives of the target audience and implementers. These data will also help provide insight into local values or concepts, barriers and facilitators to implementing what was learned in the parenting program, and an understanding of the elements that participants value in terms of reintegration. Data will be collected from focus groups and child-friendly individual activity-based approaches with reunified children from both comparison and intervention arms.

Data Management: Quantitative data will be collected by trained interviewers on Google Nexus tablets using Open Data Kit (ODK) software. Tablets will be password protected with encrypted hard drives. At the end of each data collection day, the data on each tablet will be transferred to Westat via a secure file transfer protocol (FTP).

Data Analysis A primary objective of the study is to determine whether there is an association between the parenting intervention and the six domains of reintegration among reunified children and their caregivers. The outcomes across the six outcome domains of reintegration will be summarized using mean, median, and standard deviation for continuous measures, and frequency and percentage for categorical measures, both within and across the two groups. The investigators will then conduct Analysis of Variance (ANOVA) to examine effects of participation in the parenting program on the outcome variables. In addition, based on preliminary analysis, the investigators may select covariates, and conduct Analysis of Covariance (ANCOVA). For outcome variables that are categorical, Chi-square tests will be conducted. To examine the changes over time within and across the groups, the investigators plan to conduct Generalized Linear Mixed Models (GLMM) with repeated measures at multiple time points.

For the main analysis to assess whether participation in a household-based parenting program results in higher rates of reintegration, the investigators will consider several options for the main analysis. One possibility will be to develop a scale using factor analysis to analyze the various domains that constitute reintegration. Exploratory Factor Analysis (EFA) will help us identify items that measure reintegration success conceptually, and have strong contributions to specific constructs. The investigators will use information based on EFA as well as the known conceptual framework for these domains to decide the number of factors and items in each factor. Confirmatory Factor Analysis (CFA) will then be performed to validate the factor structure developed based on findings from the EFA. Another possibility will be to conduct multivariate GLMM to form composites of the outcome variables that can be analyzed together. That is, variables within each dimension and across the dimension can be conceptualized, categorized and then entered as dependent variables in the multivariate GLMM analysis to examine the effect of the intervention on outcomes over time. The investigators will also use GLMM to examine whether the improvement in outcomes over time in the intervention group are significantly greater than the improvement in outcomes in the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* The case assessment indicates that the child can be reunified with the family/kin.
* Child is being reintegrated with family or kin in one of the study districts.

Exclusion Criteria:

* Child requires an alternative care arrangement including foster care, adoption, or independent/group home living.
* Child has severe developmental disabilities.
* Children whose caregivers plan to send them boarding school

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Increase in positive parenting behaviors (supportive positive behaviors, and setting limits) | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Positive parenting behaviors of parental involvement and setting limits will be measured by the Parenting Young Children Scale (PARYC; McEachern, Dishion, Weaver, Shaw, Wilson & Gardner, 2012). The PARYC is a measure designed to address parenting behaviors relevant for the caregivers of young children in the past month. The PARYC has been used widely including in Africa such as in South Africa as part of the Sinovuyo Teen trial (Cluver et al., 2016). It has 21 items measuring the occurrence of specific parental behavior towards children during the previous month on a 7-point Likert scale (0 = never; 6 = always). We will use subscales of Supporting Positive Behavior for children aged 1-13 years (7 items), and Setting Limits for ages 1-5 (7 items). In our study, both subscales of the PARYC will be administered to the Home and the RCF caregivers; the Supporting Positive Behavior subscale will be administered to children 8 years and above, with a modified 5-point rating scale.
Increase in positive parenting behaviors (positive involvement and monitoring/supervision) | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Positive parenting behaviors of positive involvement and monitoring/supervision will be measured using the Alabama Parenting Questionnaire (APQ; Frick 1991). The APQ has been used widely including in studies in Africa, such as in South Africa (Casale et al., 2015) and as part of the Sinovuyo Teen parenting program (Cluver et al., 2016). The APQ has 42 items related to the etiology of child externalizing problems. Respondents are asked to select how often various actions (e.g., "Your child is home without adult supervision.") happen typically on a 5-point Likert-like scale (1 = never; 5 = always). For this study, we will be using the APQ subscales of Involvement for children aged 1-13 years (10 items), and Monitoring and Supervision subscale for ages 6-13 (10 items). In our study, the APQ child form will be administered to children 8 years and older; the APQ parent form will be administered to the home and the RCF caregiver.
Increased levels of secure attachment | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Attachment behaviors of children aged 1 to 6 years will be assessed by the Disturbances in Attachment Interview (Smyke & Zeanah, 1999). This is a semi-structured interview with questions to the child's primary caregiver about the child's typical behaviors. The DAI includes 12 items - 8 questions on Disturbances of Non-attachment and 4 questions on Secure-Base distortions. Each item is explored through a series of probes. Trained interviewers rate each item as "0" = none or never, 1= somewhat or sometimes, and 2 = considerable or frequently; responses are summed with higher scores indicating greater disturbances in attachment. The DAI will be administered to the RCF caregiver at baseline, and the Home caregiver 6- and 12-months follow-up.
Decrease in Child Problem Behaviors | Baseline, 6 months post- reunification and 12-month post-reunification follow-up
  Child Problem Behaviors will be measured by the Child Behavior Checklist (CBCL, Achenbach 1992). The CBCL has been used widely including in studies in Africa, such as in South Africa as part of the Sinovuyo Teen parenting program (Cluver et al., 2016). CBCL is a caregiver-report questionnaire on which the child will be rated as either a 0 ("Not True"), 1 ("Somewhat or Sometimes True"), or a 2 ("Very True or Often True"), on various behavioral and emotional problems. It assesses internalizing (i.e., anxious, depressive, and overcontrolled) and externalizing (i.e., aggressive, hyperactive, noncompliant, and undercontrolled) behaviors. We will use the two versions, one for children aged 1 to 5 years, and another for children aged 6 to 13 years. CBCL will be rated by both the home caregiver as well as the RCF caregiver.
Better attitudes towards physical punishment in children | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Attitudes towards discipline and physical punishment will be measured by using items from the International Child Abuse Screening Tool Attitudes measure, developed for the Sinovuyo study (Cluver et al., 2016). The ICAST-Attitudes has 3 items that measure attitudes towards physical punishment of children using the example of a child who is "always getting into trouble". Respondents are asked how 'good' the disciplining tactics are using a scale of 1 ("very good") to 5 ("very bad"). The measure will be administered to the home caregiver, the RCF caregiver, and the 8+ child.
Lowered report of child abuse | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Child abuse will be measured using an abbreviated version of the International Society for the Prevention of Child Abuse and Neglect child and caregiver version of the International Child Abuse Screening Tool (Reduced ICAST-Trial). The Reduced ICAST has questions that pertains to incidents of violence in the past months. The ICAST measures three types of abuse: physical abuse, emotional abuse, and sexual abuse. In this study, the response code was adapted to a frequency scale from 0 to more than 8 times as certain behavior occurred in the past month. The Reduced ICAST will be administered to the RCF caregiver and the 8+ child. The RCF caregiver version has 14 items. The 8+ Child version has 20 items and includes questions on whether the child has asked for help relating to the questions that are not part of the ICAST tool. The investigators will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Increase in child Cognitive functioning | Baseline, 6-month post- reunification follow-up
  Cognitive functioning of younger children, aged 1 to 4 years, will be assessed by the Mullen Scales Early Learning (MSEL; Mullen, 1995). MSEL is an individually administered standardized measure of cognitive ability and motor development, which has been used in many studies in Uganda and other countries in Africa (Boivin et al., 2013). We will be administering all five scales of MSEL: Gross Motor, Fine Motor, Visual Reception, Receptive Language, and Expressive Language that are combined into an Early Learning Composite score. Raw scores will be converted to standardized score that will yield a composite of the Mental Processing Index (MPI).
  Cognitive functioning of older children, aged 5 to 13, will be assessed by the Kaufman Assessment Battery for Children (KABC-II; Kaufman & Kaufman, 2004). It is an individually administered standardized measure of sequential and simultaneous processing, learning, reasoning, and crystallized knowledge ability, which has been used in many studies
Increased access to food | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Household food security is measured at all 3 time points (in the Caregiver questionnaire) by the Household Hunger Scale (HHS, Ballard, Coates, Swindale, & Deitchler, 2011). The HHS is a series of three questions regarding household food insecurity in the prior month (i.e., "was there ever no food to eat of any kind…?" [and, if so, how often: rarely (1-2 times), sometimes (3-10 times), often (more than 10 times)]; "did you or any member of your household go to sleep at night hungry…?" [and how often]; and "did you or any household member go a whole day and night without eating anything at all because there was not enough food?" [and how often]). The HHS will be administered only to the home Caregiver at all time points.
Increased access to health care | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Children's access to health care will be measured by questions on availability of shelter and clothing, general health, schedule of immunizations, and access to medical care. These questions were based on existing OVC tools and questions used in the Sinovuyo study (Cluver et al., 2016). These questions will be administered to the RCF caregiver and the 8+ child. The schedule of immunizations will be obtained from the child's vaccination card at the RCF.
Increase in child and caregiver's Self-Esteem | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Child and the home caregiver's self-esteem will be assessed by Rosenberg Self-Esteem Scale (Rosenberg, 1965), which is a 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. All items are answered by the respondent using a 4-point Likert scale format ranging from "strongly agree" to "strongly disagree". The self-esteem scale will be administered to the Home Caregiver and the 8+ Child.
Increase in Home Caregiver's Psychosocial Health | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  The home caregiver's symptoms of psychosocial health will be assessed by The Shona Symptom Questionnaire (SSQ) that was developed in sub-Saharan Africa (Patel, Simunyu, Gwanzura, Lewis, & Mann, 1997). The SSQ consists of 14 "yes/no" questions pertaining to common symptoms of mental disorder, and idioms or distress of primary care attenders. The items are a mixture of emic and etic phenomena, and are self-rated by the respondent. The SSQ will be administered only to the Home Caregiver at all time points.
Decrease in Parenting Stress | Baseline, 6 months post- reunification and 12-month post-reunification follow-up
  Parenting stress of the home caregiver will be measured using the Parental Stress Scale (PSS; Berry & Jones, 1995). The PSS has been used widely including in studies in Africa, such as in South Africa as part of the Sinovuyo Teen parenting program (Cluver et al., 2016). PSS is a self-report scale that contains 18 items representing pleasure or positive themes of parenthood (emotional benefits, self-enrichment, personal development) and negative components (demands on resources, opportunity costs and restrictions). Respondents are asked to agree or disagree with items in terms of their typical relationship with their child or children and to rate each item on a five-point scale ranging from "strongly disagree" (1) to "strongly agree" (5). The PSS will be administered only to the Home Caregiver at all time points.
Decrease in child and caregiver's loneliness | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Home caregiver's and child's (8+ years) loneliness will be measured using UCLA Loneliness scale (Version 3, Russell, D. (1996)), designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. We will be using the 3-item scale (Hughes, Waite, Hawkley, & Cacioppo, 2004) that will be self-rated on a 4-point scale as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), or N ("I never feel this way").
Decrease in child's depressive symptoms | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Children's Depression Inventory (CDI; Kovacs, 2011) will be used to assess self-rated depressive symptoms of older children (aged 8 yrs. and above). CDI measures cognitive, affective, and behavioral symptoms of depression such as depressed mood, hedonic capacity, vegetative functions self-evaluation and interpersonal behaviors in the past two weeks. It covers the consequences of depression as they relate to children and functioning in school and with peers. We will use the 2nd edition (CDI2) with 12 items. For each item the child has three possible answers; 0 indicating an absence of symptoms, 1 indicating mild symptoms, and 2, definite symptoms.
Increase in Protective Factors and Resilience | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  The presence of a caring adult as a protective factor will be assessed using questions from the core module of The California Healthy Kids Survey (CHKS, 2014; CA Department of Education, Version H18 - Fall 2014 - Spring 2015). CHKS has been administered as a comprehensive, youth risk behavior and resilience survey . The four items pertain to child's perception of the availability of a caring adult. The items are rated on a 4-point scale: Not at all true, A little true, Pretty much true, and very much true." Of the original 6 questions, 2 questions were removed at the piloting stage. In the present study, this measure will be administered to the older children (8+ years).
Increased levels of social support for caregiver and child | Baseline, post- intervention and 12-month post-intervention follow-up
  Perceived social support will be measured using the Medical Outcome Study Social Support Questionnaire (MOS-SSQ, Sherbourne & Stewart, 1991). The MOS-SSQ has been used widely including in studies in Africa, such as in South Africa (Lachman et al., 2014) and as part of the Sinovuyo Teen parenting program (Cluver et al., 2016). The MOS-SSQ is a 19-item survey that measures emotional/informational support, tangible/instrumental support, affectionate support, and positive social interaction. Respondents report on the frequency of how often they receive support (e.g., "someone you can count on to listen to when you need to talk") on a Likert-like scale of 1 to 5 (1 = none of the time; 5 = all of the time). Total scores are calculated by averaging the scores for each item and then transformed into a 0 to 100 scale. The MOS-SSQ will be administered to the Home Caregiver and the 8+ Child.
Increased sense of community belonging for caregiver and child | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Sense of community belonging will be measured by an adapted version of the RETRAK and ASPIRE's 3-item sense of belonging feelings of acceptance and involvement in the community. ASPIRES Family Care: Longitudinal Project Assessment Research, Child Integration Status Tool, Version 2.0, 2016. The measure will be administered to the Home caregiver and the 8+ child.
School enrollment | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  School enrollment will be assessed based on self-reports. Questions on school enrollment, type of school, reasons for lack of enrollment, number of days missed, current grade, previous grade, repetition of a grade, will be asked of the RCF caregiver, home caregiver, and the 8+ child.
Satisfaction with school | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Children's and caregiver's satisfaction with child's schooling will be measured by a 3-item questionnaire; children's feeling safe at school, having a sense of belonging at school.

SECONDARY OUTCOMES:
Child Anthropometry: Height | Baseline, 6-month post- reunification and 12-month post- reunification follow-u
  Children's height (in centimeters) based on standardized measurement of the child at the RCF.
Child Anthropometry: Weight | Baseline, 6-month post- reunification and 12-month post- reunification follow-u
  Children's weight (in kilograms) based on standardized measurement of the child at the RCF.
Satisfaction of the intervention | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Satisfaction and feasibility of the intervention will be measured qualitatively. Interviews and focus groups will be conducted of the caregivers, children, parenting facilitators, and case managers. The interviews/focus groups will be audio recorded and coded to assess a) the satisfaction and feasibility of the intervention components for children and caregivers as well as the program implementers (parenting facilitators and case managers); b) effect of the individual intervention components on the reintegration process from the perspectives of the target audience and implementers, and c) barriers and facilitators to implementing the parenting program.

OTHER OUTCOMES:
Moderator: Child, home caregiver, and household characteristics | Baseline
  Basic caregiver and child demographic information will be asked using items adapted from validated instruments such as the UNICEF Multiple Indicator Cluster Surveys (MICS) and the Demographic and Health Survey (DHS), as well as the Sinovuyo questionnaires. For example, a household roster (similar to MICS and the DHS) is collected in the Caregiver baseline questionnaire, containing questions on household composition and HH members' age, sex, literacy, education level, and relationship to the child being reunified. Other household characteristics are also collected in the Caregiver baseline questionnaire, such as dwelling characteristics, household assets (similar to the household assets module in the DHS, used to measure HH wealth). We also added questions specific to the current study such as the presence of child's biological parents (including reasons for absence), reasons for living in the RCF.
Moderator: Home Caregiver's Marital Quality | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  The home caregiver's marital quality, or quality of relationship with the current partner, will be assessed using the Quality of Marriage Index (QMI, Norton, R.; 1983). The QMI is a 5-item measure of marital satisfaction. Respondents answer the items on a 7- point scale ranging from 1 (strongly disagree) to 7 (strongly agree). The QMI will be administered to home caregivers who are in a current relationship.
Moderator: Home Caregiver's exposure to Intimate partner violence | Baseline, 6-month post- reunification and 12-month post- reunification follow-u
  The home caregiver's exposure of intimate partner violence will be measured by short form of the Revised Conflict Tactics Scale (CTS2S, Straus & Douglas, 2004). The CTS2S is a 20-item measure of both the extent to which partners in a dating, cohabiting, or marital relationship engage in psychological and physical attacks on each other, and their use of reasoning or negotiation to deal with conflicts. All items are answered by the respondent using a 5-point Likert scale format ranging from "strongly disagree" to "strongly agree".
Moderator: Alcohol use in home caregivers | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  The Alcohol Use Disorders Identification Test (AUDIT) measures the use of alcoholic beverages by the caregiver (World Health Organization, Babor, Higgins-Biddle, Saunders, & Monteiro, 2001). AUDIT has been used in many studies in Africa, more recently in Lesotho (Tomlinson et al., 2016), to assess alcohol consumption and drinking behaviors. We selected three questions pertaining to the frequency of alcohol use in the past year. Used in The AUDIT will be administered to the home caregiver
Moderator: Child disability | Baseline, 6-month post- reunification and 12-month post- reunification follow-up
  Child disability will be assessed using the disability module from the UNICEF Multiple Indicator Cluster Surveys (MICS) (Cappa 2011).. The "10 Questions" (TQ) Child disability module, which was standardized in the 3rd round of MICS surveys (MICS3) in 2005-2006, uses questions posed to the parent or caregiver of children aged 2-9. These questions focus on activity limitations and participation restrictions, and they rely on observations of the caregiver of the difficulty the child may experience in seeing, hearing, walking or climbing steps, remembering, understanding and communicating in his/her usual language. Response options have been simplified to "yes" or "no" for each item.
Moderator: Caregiver's experience of abuse during childhood | Baseline
  Caregiver's experience of abuse as a child will be assessed using an adapted version of the International Society for the Prevention of Child Abuse and Neglect's Child Abuse Screening Tools - Retrospective Version (ICAST-R; Dunne, Zolotorb, Runyanb, Andreva-Millerc, Yuen, Chood, Dunnea, S., ... Youssefj, R. (2009); Lachman et al., 2017). We use the version with 7 items that was adapted for the Sinuvuyo study (Cluver et al., 2016), by selecting a subset of the items pertaining to sexual abuse with possible responses as "yes" or a "no". This scale utilizes parent self-report of experiences during their own childhood to assess the history of incidence of physical maltreatment, verbal abuse, and sexual abuse. In this study, incidence of past history of child maltreatment will be scored as dichotomous variables for physical, verbal, and sexual abuse, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse).

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Ihrig, MSW, Study Director — Catholic Relief Services
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lachman JM, Cluver L, Ward CL, Hutchings J, Mlotshwa S, Wessels I, Gardner F. Randomized controlled trial of a parenting program to reduce the risk of child maltreatment in South Africa. Child Abuse Negl. 2017 Oct;72:338-351. doi: 10.1016/j.chiabu.2017.08.014. Epub 2017 Sep 4. PMID 28881303
- [Background] Bangirana P, Opoka RO, Boivin MJ, Idro R, Hodges JS, John CC. Neurocognitive domains affected by cerebral malaria and severe malarial anemia in children. Learn Individ Differ. 2016 Feb;46:38-44. doi: 10.1016/j.lindif.2015.01.010. Epub 2015 Jan 16. PMID 27212870
- [Background] Tomlinson M, Skeen S, Marlow M, Cluver L, Cooper P, Murray L, Mofokeng S, Morley N, Makhetha M, Gordon S, Esterhuizen T, Sherr L. Improving early childhood care and development, HIV-testing, treatment and support, and nutrition in Mokhotlong, Lesotho: study protocol for a cluster randomized controlled trial. Trials. 2016 Nov 9;17(1):538. doi: 10.1186/s13063-016-1658-9. PMID 27829445
- [Background] Herrero Romero R, Hall J, Cluver L, Meinck F. Can supportive parenting protect against school delay amongst violence-exposed adolescents in South Africa? Child Abuse Negl. 2018 Apr;78:31-45. doi: 10.1016/j.chiabu.2017.09.025. Epub 2017 Sep 28. PMID 28964563